CLINICAL TRIAL: NCT01639040
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Assess the Safety of REGN668 Administered Concomitantly With Topical Corticosteroids to Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study to Assess the Safety of Dupilumab (REGN668/SAR231893) Administered Concomitantly With Topical Corticosteroids (TCS) in Patients With Moderate-to-severe Atopic Dermatitis (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1121
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo QW (Experimental): Placebo (for Dupilumab) once weekly (QW) for 4 weeks by subcutaneous injection with the background therapy of potent topical corticosteroid (TCS) for up to 28 days
  Interventions: Drug: Placebo (for Dupilumab); Other: Topical Corticosteroid (TCS)
- Dupilumab 300 mg QW (Experimental): Dupilumab 300 mg once weekly (QW) for 4 weeks by subcutaneous injection with the background therapy of potent TCS for up to 28 days
  Interventions: Drug: Dupilumab; Other: Topical Corticosteroid (TCS)

INTERVENTIONS:
Drug: Dupilumab — Dupilumab 300 mg once weekly (QW) for 4 weeks
  Other Names: REGN668; SAR231893; Dupixent
  Arms: Dupilumab 300 mg QW
Drug: Placebo (for Dupilumab) — Placebo (for Dupilumab) once weekly (QW) for 4 weeks
  Arms: Placebo QW
Other: Topical Corticosteroid (TCS) — TCS such as methylprednisolone aceponate 0.1%, mometasone furoate 0.1%, or betamethasone valerate 0.1%

SUMMARY:
The purpose of this study was to assess the safety of Dupilumab administered concomitantly with topical corticosteroids (TCS) in patients with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or older
2. Chronic AD that had been present for at least 2 years

Exclusion Criteria:

1. Prior treatment with Dupilumab
2. Hypersensitivity to corticosteroids or to any other ingredients contained by the TCS product used in the study
3. AD lesions located on face, flexural, and genital areas
4. Certain treatments and medical procedures, undertaken within a particular time frame prior to the baseline visit, preclude eligibility for participation in the study
5. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit
6. Treatment with an investigational drug within 8 weeks
7. Known history of human immunodeficiency virus (HIV) infection
8. Presence of certain laboratory abnormalities at the screening visit
9. History of certain opportunistic infections or certain clinical parasite infections
10. History of malignancy within 5 years before the baseline visit, with certain exceptions
11. Pregnant or breast-feeding women
12. Travel within 12 months of study start to areas endemic for parasitic infections, such as developing countries in Africa and the tropical and subtropical regions of Asia
13. History of alcohol or drug abuse within 2 years of the screening visit
14. Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the patient at risk, interfere with participation in the study, or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (13):
- Germany (7):
  - Berlin
  - Dresden
  - Dülmen
  - Frankfurt
  - Gera
  - Langenau
  - Münster
- Hungary (2):
  - Szeged-Hungary
  - Szolnok
- Poland (4):
  - Gdansk
  - Lodz
  - Lublin
  - Warsaw

REFERENCES:
- [Result] Beck LA, Thaci D, Hamilton JD, Graham NM, Bieber T, Rocklin R, Ming JE, Ren H, Kao R, Simpson E, Ardeleanu M, Weinstein SP, Pirozzi G, Guttman-Yassky E, Suarez-Farinas M, Hager MD, Stahl N, Yancopoulos GD, Radin AR. Dupilumab treatment in adults with moderate-to-severe atopic dermatitis. N Engl J Med. 2014 Jul 10;371(2):130-9. doi: 10.1056/NEJMoa1314768. PMID 25006719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 participants were screened in the study between 30 July 2012 and 20 December 2012.
Pre-assignment Details: Out of 38 participants, 31 were randomized and treated in the study. Participants were randomized in 2:1 ratio to receive Dupilumab 300 mg or Placebo.
Period: Overall Study
Arm/Group | Placebo QW | Dupilumab 300 mg QW
Started | 10 | 21
Completed | 9 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo (for REGN668) once weekly for 4 weeks by subcutaneous injection with the background therapy of potent TCS for up to 28 days.
- REGN668 300 mg: REGN668 300 mg once weekly for 4 weeks by subcutaneous injection with the background therapy of potent TCS for up to 28 days
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN668 300 mg | Total
Number analyzed (Participants) | 10 | 21 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (16.73) | 36.0 (11.26) | 36.6 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 5 | 8 | 13
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  units on a scale | 24.1 (12.70) | 23.1 (12.35) | 23.4 (12.26)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 6-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe; and 5 = very severe disease) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  units on a scale | 3.4 (0.47) | 3.4 (0.60) | 3.4 (0.55)
Pruritus Numerical Rating Scale (NRS) score [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS was an assessment tool that was used to report intensity of subject's pruritus (itch), both maximum and average intensity during a 24-hour recall period. Participants were asked following question: how would a subject rate his itch at worst moment during previous 24 hours (for maximum itch intensity on a scale of 0-10 [0 = no itch; 10 = worst itch imaginable]).
  units on a scale | 5.0 (1.39) | 6.4 (2.00) | 6.0 (1.93)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a subject who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on-treatment period (from start of administration of first dose of study drug to the end of study [up to Day 78]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline up to the end of study (up to Day 78)
Population: Safety population included all randomized participants who received any study drug; based on the treatment received (as treated).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg QW
Number analyzed (Participants) | 10 | 21
percentage of participants
  With at least one TEAE | 70.0 | 57.1
  With study drug related TEAEs | 40.0 | 28.6
  With serious TEAEs | 10.0 | 0
  With TEAEs resulting in study discontinuation | 10.0 | 0

2. Other Pre Specified Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Score: Reduction of ≥50 at Day 29 - Censored Last Observation Carried Forward (LOCF)
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. The efficacy data were set to missing after prohibited medication was used or after the participant was discontinued from the study. Then, all missing values were imputed by simple LOCF.
Time Frame: Day 29
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline assessment; it was based on the treatment allocated (as randomized).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg QW
Number analyzed (Participants) | 10 | 21
percentage of participants | 50.0 [18.7 to 81.3] | 100.0 [83.9 to 100.0]

3. Other Pre Specified Outcome: Percent Change in Pruritus Numerical Rating Scale (NRS) From Day 1 (Baseline) to Day 29 (Week 4)
Description: Pruritus NRS was an assessment tool that was used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).
Time Frame: Baseline up to Day 29
Population: FAS included all randomized participants who received at least 1 dose of study medication and had at least 1 post-baseline assessment; it was based on the treatment allocated (as randomized).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | REGN668 300 mg
Number analyzed (Participants) | 10 | 21
percent change | -24.7 (47.30) | -70.7 (21.45)

4. Other Pre Specified Outcome: Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of "0" or "1" at Day 29
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
Time Frame: Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | REGN668 300 mg
Number analyzed (Participants) | 10 | 21
percentage of participants | 30.0 [6.7 to 65.2] | 52.4 [29.8 to 74.3]

5. Other Pre Specified Outcome: Percent Change in Investigator's Global Assessment (IGA) Score From Day 1 (Baseline) to Day 29 (Week 4) - Censored LOCF
Description: IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear). The efficacy data were set to missing after prohibited medication was used or after the participant was discontinued from the study. Then, all missing values were imputed by simple LOCF.
Time Frame: Baseline up to Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | REGN668 300 mg
Number analyzed (Participants) | 10 | 21
percent change | -30.6 (39.00) | -52.5 (21.44)

6. Other Pre Specified Outcome: Percent Change in Eczema Area and Severity Index (EASI) Score From Day 1 (Baseline) to Day 29 (Week 4) - Censored LOCF
Description: EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. The efficacy data were set to missing after prohibited medication was used or after the participant was discontinued from the study. Then, all missing values were imputed by simple LOCF.
Time Frame: Baseline up to Day 29
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent Change
Arm/Group | Placebo | REGN668 300 mg
Number analyzed (Participants) | 10 | 21
percent Change | -52.5 (39.53) | -75.6 (13.29)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 78) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (day from first dose of study drug to the end of study visit [up to Day 78]).
Arm/Group | Placebo | REGN668 300 mg
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/21
Other Adverse Events (participants affected / at risk) | 7/10 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | REGN668 300 mg (N=21)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | REGN668 300 mg (N=21)
Injection site erythema (General disorders) | 1 (4) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (6)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (6) | 3 (8)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)

LIMITATIONS AND CAVEATS:
This was a small safety study that was not adequately powered to assess efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.